CLINICAL TRIAL: NCT06627114
Title: Effectiveness of Nutrition Education Program and Omega-3 Supplementation on Body Weight, Liver Enzymes, Lipid Profile Among Non-Alcoholic Fatty Liver Disease Patients
Brief Title: Effectiveness of Nutrition Education Program and Omega-3 Supplementation Among Non-alcoholic Fatty Liver Disease Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Dilkhosh Shamal Ramadhan, lecturer, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nutrition education VS Omega-3
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Omega-3 Supplementation; Nutrition Education Program
Keywords: Nutrition Education; Omega-3 Supplementation; Body Weight; Liver Enzyme; Lipid Profile; Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Body Weight | interventions — Fatty Acids, Omega-3; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nutrition education Program (Active Comparator): patients randomized to the intervention group, will participate in a nutritional education. the nutrition education sessions will be based on theory of planned behavior, which will include three 45-60-minute sessions about understanding NAFLD and nutrition basics, the role of social influences and support systems in managing NAFLD and overcoming barriers and building confidence.
  Several educational methods will be using such as lectures, slides, group discussion, question and answers, instructional images, poster, booklet and Use case studies or scenarios. Participants will encourage to increase the intake of fruits, vegetables, complex carbohydrate, low fat dairy, healthy fats, white meat and fish, and also avoid the intake of unhealthy fats and refined carbohydrates. Furthermore, in each session, will be reviewing the patients' dietary practice and provided recommendations. Adherence to dietary intervention will assess by weekly phone calls and dietary records.
  Interventions: Behavioral: nutrition education program
- Omega-3 supplementation (Active Comparator): Omega-3 Arm:1000 mg omega-3 fatty acids soft gel capsules (containing DHA 220 mg and EPA 330 mg) in two dose per day, to be taken orally with meal. Planned duration of the treatment is 12 weeks.
  Interventions: Dietary Supplement: Omega 3 fatty acids
- control (Active Comparator): Patients randomized to the control group, who receive routine care at the outpatient clinic in Rizgari teaching hospital. At baseline, a physician will explain the laboratory test results and the natural history of NAFLD to the patients.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: nutrition education program — Nutritional Guidance: Emphasizing a balanced diet rich in fruits, vegetables, whole grains, lean proteins, and healthy fats while reducing processed foods, sugars, and saturated fats.
  Weight Management: Encouraging gradual weight loss if overweight, as this can significantly improve liver health.
  Individualized Plans: Tailoring nutrition education to the individual needs, preferences, and any other underlying health conditions.
  Monitoring and Support: Providing ongoing support and education to help participants make sustainable changes and track their progress.
  Arms: Nutrition education Program
Dietary Supplement: Omega 3 fatty acids — Omega-3 Arm:1000 mg omega-3 fatty acids soft gel capsules twice daily, to be taken orally with meal.
  Arms: Omega-3 supplementation
Other: control group — receive routine care at the outpatient clinic. At baseline, a physician will explain the laboratory test results and the natural history of NAFLD to the patients.
  Arms: control

SUMMARY:
The aim of this clinical trial is to examine the impact of nutritional education and omega-3 supplementation in influencing body weight, liver enzyme levels, and lipid profiles in patients diagnosed with non-alcoholic fatty liver disease.

Eligible patients who have non-alcoholic fatty liver disease are randomized to receive either nutritional education, omega-3 fatty acids containing DHA and EPA, or control groups.

the main questions are: Does the Nutrition education affect body mass, liver enzyme and lipid profile in patient with non-alcoholic fatty liver disease? Does Omega-3 supplementation affect body mass, liver enzyme and lipid profile in patient with non-alcoholic fatty liver disease?

The expected outcome will improvement in the laboratory liver tests, liver steatosis on ultrasound, and lipid profile and also decrease body weight.

DETAILED DESCRIPTION:
159 participants with non-alcoholic fatty liver disease patient who will attend Rizgary Teaching Hospital in Erbil City.

In order to obtain the accurate data and representative sample, Eligible patients will be randomized to one of three arms:

1. those who will receive nutritional education (For nutritional education intervention, Theory of planned behavior-based interventions for the non-alcoholic fatty liver disease patients will include three educational sessions).
2. those who will receive omega-3 supplements (the dose of omega-3 (DHA+ EPA) will be 1000 mg twice daily).

   or
3. to a control group who will not receive any intervention, (who receive routine care at the outpatient clinic).

Data collection will depend on face-to-face interviews including baseline, using validated questionnaires, ultrasonography and laboratory test (liver enzyme and lipid profile) at first visit, mid and after 12 weeks of intervention.

Tools for data collection The questionnaire that will be developed for the purpose of data collection. Data will collect through using the questionnaire that consisted of the following parts: Baseline characteristics of the study participants. such as (name, age, sex, marital status, level of education, occupation, mobile number, body mass index), and theory of planned behavior will construct (TPB) who will receive nutritional education intervention, for a NAFLD diagnosis, ultrasound proof of fatty liver (stage I or above) and biochemical parameter such as an elevated level of liver enzymes will require. An experienced radiologist will do the ultrasonography. The grade of fatty liver will determine based on hepatic parenchymal brightness by ultrasound, and established methods will use to test the liver's biochemical parameters such as lipid profile (cholesterol LDL, cholesterol HDL, Triglycerides, and Total cholesterol). and liver AST, ALT, ALP and GGT). And measuring body mass index will be measure at the baseline and after 12-weeks of intervention among NAFLD patients who will receive either nutritional education, omega-3 supplementation and control group. The questionnaire will modify based on the literature review and feedback of experts, which is applicable and specific to the study also translated to Kurdish language.

The validity of the study:

Tools will be designed by the researcher after reviewing the relevant literature and tested for its content validity. The questionnaire will be sent to panel of experts from different health specialty (such as Community health nursing, hepatologist medicine, community medicine specialist) to assess the relevance of tool with title and objectives. The responses will be represented in four points score ranging from (4-1); 4= strongly relevant, 3= relevant, 2= little relevant, and 1= not relevant by use Liker scale.

The Reliability of the study:

Consistency of questionnaire will be tested by Cronbach's alpha test (test-re-test) reliability will be checked on that answered the questionnaire twice. A correlation analysis will be performed on the scores of the two tests (observations test and knowledge test), Test-Retest will be done by 10non alcoholic fatty liver disease patients who will not part of the samples.

Pilot study:

The pilot study will be carried out on 10 non- alcoholic fatty liver disease patients to test all tools for clarity, objectivity, relevance, feasibility and the applicability of the tools. It also will conduct to identify any problem associated with administering the tools and measure the time needed for data collection then the necessary modifications will be conducted accordingly. Data included in pilot study will be excluded from the current study.

Implementation of the interventional program:

The interventional program will focus on nutrition education and omega-3 supplementation ways, which was implemented through the sessions. The nutritional interventional program sessions were administrated individually or in small group and each session was designed and scheduled for approximately45-60 minutes.

First phase: an interview session The researcher will introduce herself to the NAFLD patients and explained the nature of the subject area to the approached ones who run across the inclusion criteria and agreed to take part in the study, then will start. The researcher will interview NAFLD patients. The NAFLD patients become aware of keeping confidentiality of information and they complete the basic information forms which will prepare by the researcher. According to Randomization criteria the NAFLD patients will be divide into two groups of intervention and one control.

Second Phase: Pre- test Pre-test assessment of each NAFLD patients in program according of each three group will expose to the pre-test questionnaire (both knowledge and lifestyle), BMI measures, Laboratory test (liver function test and lipid profile).

Third Phase: Intervention among NAFLD patients The Intervention among NAFLD patients. According to Randomization criteria the NAFLD patients will be divide into three groups, two groups of intervention and one control. In nutrition education group, will interview individually or in small groups.

Fourth Phase: Post- Test After 12 weeks of the completion, the posttest will administer to collect knowledge and changes of daily life for all NAFLD patients and referring them for ultrasound and making laboratory test liver enzyme such as (AST, ALT, ALP and GGTP) and lipid profile such as (cholesterol LDL, cholesterol HDL, Triglycerides, and Total cholesterol) in three groups will do.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-74 years' old.
* Ability to use a mobile phone.
* Ultrasound examination diagnosed Patients with grade 1 and 2 non-alcoholic fatty liver disease.

Exclusion Criteria:

* supplementary intakes of n-3 PUFA within the previous 6 months.
* pregnancy or breastfeeding.
* chronic liver disease of other causes (autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, hereditary haemochromatosis, Wilson's disease, a1-anti-trypsin deficiency, coeliac disease).
* hormone therapy and use of drugs like amiodarone, methotrexate, and corticosteroid.
* three months.
* chronic disease such as cardiovascular, gastrointestinal, thyroid, renal, cancer or pancreatic that assessed by a specialist.
* The use of drugs known to be associated with liver steatosis (Drugs known to be capable of inducing steatosis and steatohepatitis can be divided into three broad groups: those that cause steatosis and steatohepatitis independently (e.g., amiodarone, perhexiline maleate); drugs which can precipitate latent NASH (e.g., tamoxifen); drugs which induce sporadic events of steatosis/steatohepatitis (e.g., carbamazepine).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Comparision the effectiveness of nutrition education and Omega-3 supplementation on reduction in hepatic steatosis scores. | hepatic steatosis scores the measurement will be taken at the baseline and through study completion, an average of 12 weeks.
  The first primary outcome measures will be the reduction in hepatic steatosis scores, will be assess by using ultrasound. The diagnosis of fatty liver will be based on parenchymal brightness, liver-to-kidney contrast, bright vessel walls, gallbladder wall definition, and diaphragmatic definition.
  The fatty disease will be graded and labeled as mild, moderate, or severe, or grades 0 to 3 (with 0 being normal) based on the degree of parenchymal brightness.
  Grade 0 (normal liver): the liver and renal cortex are of similar echogenicity. Grade 1 (mild): slight diffuse increase in the fine echoes of liver parenchyma with appreciable periportal and diaphragmatic echogenicity.
  Grade 2 (moderate): moderately diffuse increase in fine echoes of the liver parenchyma obscuring periportal echogenicity, but diaphragmatic echogenicity is still appreciable.
Comparision the effectiveness of nutrition education and Omega-3 supplementation on changes in serum concentrations of liver enzymes. | liver enzymes measurement will be taken at the baseline and through study completion, an average of 12 weeks.
  Description: The second primary outcome measures will be the changes in serum concentrations of liver enzymes (AST, ALT, ALP and GGT). Established methods will use to test the liver's biochemical parameters, that will be measure through using enzymatic colorimetric assays.
Comparision the effectiveness of nutrition education and Omega-3 supplementation on changes in serum concentrations of lipid profile. | lipid profile measurement will be taken at the baseline and through study completion, an average of 12 weeks.
  Description: The third primary outcome measures will be the changes in serum concentrations of lipid profile (Triglycerides, Total cholesterol, LDL-c and HDL-c). Serum TG, TC, HDL-c will be determined by enzymatic colorimetric assay method. The Friedewald formula has long been used to calculate LDL-c from total cholesterol, triglyceride, and HDL-c .

SECONDARY OUTCOMES:
comparison the effectiveness of nutrition education and omega-3 supplementation on changes in body weight measurements. | the time frame of the body weight measurement from baseline to through study completion, an average of 12 weeks.
  The first secondary outcomes were changes in body weight, among non-alcoholic fatty liver disease patients.
  body weight: measures by a calibrate digital scale. will be measure barefoot and in light clothing to the nearest 0.5 kg using a reliable scale (Seca).
comparison the effectiveness of nutrition education and omega-3 supplementation on changes in waist circumference measurements. | the time frame of the waist circumference measurement from baseline to through study completion, an average of 12 weeks.
  The second secondary outcomes were changes waist circumferences among non-alcoholic fatty liver disease patients.
  waist circumferences: use a flexible tape measure, in which in a standing position. Wrap a tape measure around your waist - it should sit right above your hip bone. Check that the tape is parallel to the floor, forming a horizontal line across your body. The tape shouldn't press into your skin, but it should be a snug fit. Take the measurement after breathing out.
comparison the effectiveness of nutrition education and omega-3 supplementation on changes in Body mass index measurements. | the time frame of the BMI measurement from baseline to through study completion, an average of 12 weeks.
  The third secondary outcomes will be changes in BMI measurements among non-alcoholic fatty liver disease patients.
  BMI: by calculation: by Measure your weight in kilograms (kg), Measure your height in meters (m). Then divide your weight by your height squared (kg/m²).
  The resulting number is your BMI.

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University, Erbil, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arab A, Hadi A, Moosavian SP, Rafie N, Hajianfar H. The Effect of Nutrition Education Program on Overweight/Obese Patients with Non-Alcoholic Fatty Liver Disease: a Single-Blind Parallel Randomized Controlled Trial. Clin Nutr Res. 2019 Jul 29;8(3):238-246. doi: 10.7762/cnr.2019.8.3.238. eCollection 2019 Jul. PMID 31384602
- [Background] Fateh HL, Rashid SA, Muhammad SS, Al-Jaf SH, Ali AM. Comparing effects of beetroot juice and Mediterranean diet on liver enzymes and sonographic appearance in patients with non-alcoholic fatty liver disease: a randomized control trials. Front Nutr. 2023 Aug 17;10:1181706. doi: 10.3389/fnut.2023.1181706. eCollection 2023. PMID 37662597
- [Background] Yan JH, Guan BJ, Gao HY, Peng XE. Omega-3 polyunsaturated fatty acid supplementation and non-alcoholic fatty liver disease: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Sep;97(37):e12271. doi: 10.1097/MD.0000000000012271. PMID 30212963
- [Background] Angelidi AM, Papadaki A, Nolen-Doerr E, Boutari C, Mantzoros CS. The effect of dietary patterns on non-alcoholic fatty liver disease diagnosed by biopsy or magnetic resonance in adults: a systematic review of randomised controlled trials. Metabolism. 2022 Apr;129:155136. doi: 10.1016/j.metabol.2022.155136. Epub 2022 Jan 13. PMID 35032545
- See also: Related Info — https://doi.org/10.7762%2Fcnr.2019.8.3.238